CLINICAL TRIAL: NCT02844556
Title: International Multicenter Study on Small Incision Lenticule Extraction(SMILE) Surgery
Brief Title: International Multicenter Study on SMILE Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Eye Hospital (Other)
Collaborators: Nethradhama Superspeciality Eye Hospital (Other); Alexandria University (Other); Belgian Ocular Laser Centre (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Jinan Mingshui Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tianjin EH-SMILE
Record Dates: First submitted 2016-07-12; First posted 2016-07-26 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Refractive Error
Keywords: SMILE surgery; FS-LASIK surgery; multicenter
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SMILE surgery (Other): Small incision lenticule extraction (SMILE) has become a novel and effective method for the correction of myopia and myopic astigmatism. It is a micro-invasive and flapless refractive procedure that has been proved to offer many advantages in terms of visual acuity, corneal sensitivity and corneal biomechanics compared with traditional refractive surgeries.
  Interventions: Procedure: SMILE surgery
- FS-LASIK surgery (Other): FS-LASIK surgery is femtosecond laser assisted- conventional refractive surgery and has also been proved to offer many advantages in terms of visual acuity, corneal sensitivity and corneal biomechanics compared with traditional refractive surgeries.
  Interventions: Other: FS-LASIK surgery

INTERVENTIONS:
Procedure: SMILE surgery — SMILE surgery and FS-LASIK surgery are both effective method for the correction of myopia and myopic astigmatism. They have been proved to offer many advantages in terms of visual acuity, corneal sensitivity and corneal biomechanics compared with traditional refractive surgeries.
  Arms: SMILE surgery
Other: FS-LASIK surgery — SMILE surgery and FS-LASIK surgery are both effective method for the correction of myopia and myopic astigmatism. They have been proved to offer many advantages in terms of visual acuity, corneal sensitivity and corneal biomechanics compared with traditional refractive surgeries.
  Arms: FS-LASIK surgery

SUMMARY:
The purpose of this study is to carry out an international multicenter trial to get more convincing and valuable results of the SMILE surgery and compare the outcomes between the SMILE surgery and the FS-LASIK (femtosecond laser assisted-laser in situ keratomileusis) surgery.

The investigators hope to investigate the differences between the SMILE and the FS-LASIK surgery comprehensively, including the comparison of visual acuity, refraction, the correction of cylindrical diopter, the high order aberrations, the corneal biomechanics, the corneal ectasia, the characteristics of the changes of central corneal thickness and the complications. To meet the demands of a multi center trial, all the examination equipments should be same in each center, and this will limit the variations within a study

DETAILED DESCRIPTION:
Hypothesis: To compare the novel refractive surgery (SMILE, the intervention group) with traditional refractive surgery (FS-LASIK, the control group) in terms of visual acuity, the higher order aberrations, corneal biomechanical parameters and the complications. SMILE surgery might offer some advantages in some aspects compared with FS-LASIK surgery.

Study program

The procedures of the study are listed as follows:

All the participants accept the refractive surgery which were selected at first, and patients' routine postoperative examinations included UCVA, BCVA, slit lamp microscopy, non-contact IOP, corneal topography with the Scheimpflug tomography system, ocular higher order aberrations using the WASCA analyzer (Carl Zeiss Meditec AG), corneal biomechanical properties acquired by the Ocular Response Analyzer and/or the Corvis ST (Corvis ST, OCULUS, Wetzlar, Germany) at 1 week, 1 month, 3 months and 6 months follow-up periods after surgery.

Statistics:

Patients who have decided to choose the SMILE surgery or the FS-LASIK will be selected as participants. The propensity matching method will be used to choose proper cases for the two groups. The propensity matching method can be calculated by SPSS software. The independent variables include: the central corneal thickness (CCT), the Km (mean Pentacam keratometry), the spherical diopter (from manifest refraction), and the cylindrical diopter (from manifest refraction), the UCVA, the BCVA, the corneal resistance factor (CRF) and the corneal hysteresis (CH) (if the investigator have the Ocular Response Analyzer) of the cornea at preoperative. The closest score of eyes in the two groups will be matched.

The data will be preserved by each site, and will be systematically collected and analyzed by TianjinEH center. The statistical expert Dr Hayes from American Pacific University will be the statistical consultant, and will also in charge of the sample size calculation, the instructor of statistical analysis, and the quality control.

ELIGIBILITY:
Inclusion Criteria:

* be accompanied by a parent or guardian who is able to give informed consent as demonstrated by signing a record of informed consent;
* at baseline, be within the age range of 18 to 45 years old inclusive
* normal corneal morphology with no corneal nebula or corneal macula, the range of preoperative K2 (the steep curvature of the 3mm area at the center of cornea) from 38.0 to 47.0 diopter
* manifest spherical equivalent of -1.0 to -10.0 diopters (D)
* cylindrical diopter no more than -5.0D
* refractive diopter maintained stable for more than2 years
* preoperative BCVA≥0.8, and the scotopic pupil diameter≥5.0mm when measured by WASCA analyzer (Carl Zeiss Meditec AG)
* picked off soft contact lens for more than 2 weeks
* picked off RGP for more than 1 month
* preoperative corneal central thickness measured by Pentacam >500μm, non-contact IOP<21mmHg
* be willing to comply with the clinical trial visit schedule as directed by the investigator.

Exclusion Criteria:

* any corneal diseases, corneal operations, eyes trauma or systemic diseases history; keratoconus or tendency of keratoconus
* corneal macula and obvious pannus; current enrolment in another clinical trial/research project.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1000 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
corrected visual acuity | change from baseline with EDTRS chart at 6 months

SECONDARY OUTCOMES:
uncorrected visual acuity | change from baseline with EDTRS chart at 6 months
spherical diopter | change from baseline with manifest refraction at 6 months
cylindrical dioptor | change from baseline with manifest refraction at 6 months
central corneal thickness | change from baseline with the Pentacam system at 6 months
corneal curvature assessed by the Pentacam system | change from baseline with mean Pentacam keratometry at 6 months
corneal resistance factor assessed by the Ocular Response Analyzer | change from baseline at 6 months
corneal hysteresis assessed by the Ocular Response Analyzer | change from baseline at 6 months
deformation amplitude assessed by the Corvis ST system | change from baseline at 6 months
spherical aberration | change from baseline with the WASCA system at 6 months
coma aberration | change from baseline with the WASCA system at 6 months
complication | intraoperative and postoperative at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wang, director, Study Director — Tianjin Eye Hospital; Sri Ganesh, professor, Principal Investigator — Nethradhama Superspeciality Eye Hospital; Bernard Heintz, professor, Principal Investigator — Belgian Ocular Laser Centre; Osama Ibrahim, professor, Principal Investigator — Cornea Center, Alexandria University; Keming Yu, professor, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Yulin Lei, professor, Principal Investigator — Jinan Mingshui Eye Hospital
Locations (1):
- Tianjin Eye Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wei S, Wang Y. Comparison of corneal sensitivity between FS-LASIK and femtosecond lenticule extraction (ReLEx flex) or small-incision lenticule extraction (ReLEx smile) for myopic eyes. Graefes Arch Clin Exp Ophthalmol. 2013 Jun;251(6):1645-54. doi: 10.1007/s00417-013-2272-0. Epub 2013 Feb 7. PMID 23389552
- [Background] Wang Y, Bao XL, Tang X, Zuo T, Geng WL, Jin Y. [Clinical study of femtosecond laser corneal small incision lenticule extraction for correction of myopia and myopic astigmatism]. Zhonghua Yan Ke Za Zhi. 2013 Apr;49(4):292-8. Chinese. PMID 23900086
- [Background] Wu D, Wang Y, Zhang L, Wei S, Tang X. Corneal biomechanical effects: small-incision lenticule extraction versus femtosecond laser-assisted laser in situ keratomileusis. J Cataract Refract Surg. 2014 Jun;40(6):954-62. doi: 10.1016/j.jcrs.2013.07.056. Epub 2014 Apr 18. PMID 24751146
- [Background] Li X, Wang Y, Dou R. Aberration compensation between anterior and posterior corneal surfaces after Small incision lenticule extraction and Femtosecond laser-assisted laser in-situ keratomileusis. Ophthalmic Physiol Opt. 2015 Sep;35(5):540-51. doi: 10.1111/opo.12226. Epub 2015 Jun 18. PMID 26087672
- [Background] Zhang J, Wang Y, Wu W, Xu L, Li X, Dou R. Vector analysis of low to moderate astigmatism with small incision lenticule extraction (SMILE): results of a 1-year follow-up. BMC Ophthalmol. 2015 Jan 24;15:8. doi: 10.1186/1471-2415-15-8. PMID 25618419